CLINICAL TRIAL: NCT06178003
Title: A Phase I/II Clinical Study of the Safety and Efficacy of Intravitreal Injection of Tpdelansbsalbac in the Treatment of Malignant Pleural and Abdominal Effusions
Brief Title: the Safety and Efficacy of Intravitreal Injection of Tpdelansbsalbac in Malignant Effusions.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHASE 003
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2023-12

CONDITIONS: Salmonella Bacteremia
Keywords: malignant pleural and abdominal effusions; Salmonella Bacteremia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intravitreal injection of Tpdelansbsalbac in malignant pleural and abdominal effusions (Experimental): the safety and efficacy of intravitreal injection of Tpdelansbsalbac in the treatment of malignant pleural and abdominal effusions
  Interventions: Biological: Tpdelansbsalbac

INTERVENTIONS:
Biological: Tpdelansbsalbac — Tpdelansbsalbac,which is Knockdown of ansB, a gene that expresses L-mentholase secreted into the extracellular region, on the basis of the genetic background of bacterium VNP20009, and construction of an ansB gene-deficient mutant strain, ΔansB.

SUMMARY:
This is a Phase I/II, open, first-in-human (FIH) study of Transebacillus in Patients with malignant pleural and abdominal effusions. It consists of Phase Ia to determine the Maximum tolerated dose (MTD) or Recommended Phase 2 dose (RP2D) of Transebacillus, and Phase Ib/II to explore and confirm the efficacy, safety and Tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate, sign the informed consent, and good compliance, able to cooperate with the diagnosis and treatment and follow-up;
* Age ≥18 years old (inclusive), male and female are not limited;
* Malignant solid tumors other than primary hepatocellular carcinoma confirmed by pathological histological or cytological examination;
* Malignant thoracic/abdominal effusion patients who have failed at least one standard antitumor systemic therapy, are not suitable for standard systemic therapy, or have no standard systemic therapy. The pleural/abdominal effusion needs to be confirmed pathologically (malignant cells found in the cytosol or pathological changes of malignancy observed in the pleural/peritoneal biopsy tissue) or clinically diagnosed as malignant pleural/abdominal effusion;
* A pleural/peritoneal effusion of intermediate or greater volume confirmed by ultrasound, which in clinical judgment requires localized treatment of the pleural/ peritoneal effusion; definition of intermediate or greater volume: maximum depth of pleural effusion ≥ 3 cm by ultrasound in sitting position; or maximum depth of abdominal effusion ≥ 4 cm by ultrasound in lying position;
* KPS score ≥ 60;
* Expected survival ≥ 3 months;
* Major organ function is essentially normal and laboratory tests；
* Screening female subjects of childbearing potential with a negative serum pregnancy test; female/male subjects of childbearing potential must be willing to use a reliable method of contraception throughout the study period (i.e., from the time of signed informed consent to 90 days after the last dose of study medication), including, but not limited to, abstinence, a male partner who has undergone a vasectomy, female sterilization, an effective intrauterine device, and effective contraceptives.
* Patients are willing to participate in the study, sign an informed consent form, and have good compliance.

Exclusion Criteria:

* Participating in or has participated in another clinical trial with investigational therapy within 4 weeks prior to first dose, or has participated in a device clinical trial within 4 weeks;
* has received systemic antitumor therapy or a drug in the thoracic-abdominal cavity within 14 days of the first intratumoral administration;
* less than 4 weeks since the need for re-puncture/drainage due to progression of the effusion after having received intraluminal therapy with cisplatin and/or an anti-angiogenic drug (e.g., Endo, bevacizumab, etc.) for the thoracic-abdominal effusion that is the subject of the treatment planned for this study;
* Has not recovered from any intervention-induced adverse event ≤ Grade 1 (except for hair loss, hearing impairment, and neurologic or endocrine disorders ≤ Grade 2 requiring replacement therapy) prior to the first dose;
* Subjects who have undergone a medium to major surgical procedure other than diagnostic or biopsy within 28 days prior to the first dose, or who are expected to undergo a major surgical procedure during the study period;
* Bilateral pleural effusion (for patients with pleural effusion) or concomitant thoracoabdominal effusion (non-enrolled treatment cavities that have not reached a moderate volume of effusion and, in the judgment of the investigator, are in stable condition and do not require clinical management may be considered for enrollment), or pericardial effusion (more than a moderate volume or with associated symptoms that, in the judgment of the investigator, require treatment) or an encapsulated effusion or celiac disease on the side of the planned treatment or have undergone within 14 days prior to the first administration of the study medication Therapeutic puncture and/or drainage (presence of suspected symptoms of effusion as well as previous history of effusion, B-ultrasound is required during the Screening Period to confirm the amount of effusion in the non-enrolled treatment cavity);
* Comorbid severe chronic obstructive pulmonary disease (global initiative for chronic obstructive lung disease (GOLD) ≥ 3), intestinal adhesions within 6 months prior to the first dose (except in patients with pleural effusions in the treatment cavity) or intestinal obstruction within 6 months prior to the first dose. Bowel obstruction within 6 months prior to the first dose;
* Severe cardiovascular disease such as New York Heart Association (NYHA) heart disease (Class III rating or better) or myocardial infarction within 6 months or current unstable angina pectoris or uncontrolled hypertension (systolic blood pressure greater than 150 mmHg and/or diastolic blood pressure greater than 100 mmHg);
* Patients with uncontrolled primary brain tumors or CNS metastases with significant intracranial hypertension or neuropsychiatric symptoms;
* Presence of uncontrolled neuropsychiatric disease, psychiatric disorders, or substance abuse that may affect compliance with the trial;
* The presence of an uncontrollable neuropsychiatric disease, psychiatric disorder, or substance abuse that may interfere with trial compliance;
* Presence of an active infection requiring systemic therapy;
* A known history of human immunodeficiency virus (HIV) infection;
* Hepatitis B virus-infected patients (HBsAg-positive or HBcAb-positive with HBV-DNA ≥2000 IU/mL or HBV-DNA ≥104 copies/mL), or Hepatitis C virus-infected patients (HCV antibody-positive with HCV-RNA quantitative test results greater than the lower limit of detection); Note: For HBV-DNA <2000 IU/mL Note: Hepatitis B virus-infected patients with HBV-DNA <2000 IU/mL or HBV DNA <104 copies/mL may be enrolled if they are willing to be treated with entecavir, tenofovir, or other antiviral therapy during the study period based on clinical judgment;
* Individuals who are allergic to any active or inactive ingredient of entrectal or co-administered chemotherapeutic agents;
* Pregnant or lactating female patients;
* Use of antibiotic drugs with caution;
* Presence of medical history or disease, therapeutic or laboratory abnormality that has the potential to interfere with the results of the trial, to prevent the subject from participating in the study in its entirety, or where participation in the study is not, in the opinion of the investigator, in the best interest of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2024-02-11 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse event (AE) | 1 months
  Laboratory tests (blood routine test, infectious markers), electrocardiogram (ECG), echocardiogram (ECHO), Physical findings, changes in vital signs.
Puncture /drainage-Free Survival (PuFS) | 1 year
  Puncture /drainage-Free Survival (PuFS) was used as an index to evaluate the efficacy of intrathecal injection in the treatment of malignant pleural or abdominal effusions.

SECONDARY OUTCOMES:
Phase Ia-Puncture /drainage-Free Survival (PuFS) | 1 year
  which was used as an index to evaluate the efficacy of intrathecal injection in the treatment of malignant pleural or abdominal effusions.
Phase Ib/II-Overall survival (OS) | 1 year
  the survival benefit of intravitreal injection of Transebacillus for the treatment of malignant thoracic or abdominal effusions as measured by overall survival
Objective remission rate (ORR) of pleural or abdominal effusion; | 1 month
  the objective remission rate of thoracic and abdominal effusions, the rate of no puncture and/or drainage at 3 months, and the time to next puncture and/or drainage (TTNP), as evaluated by the WHO Efficacy Criteria for Thoracic and Abdominal Fluids;
Time to next puncture and/or drainage (TTNP); | 1 year
  the change in symptoms and quality of life of subjects treated with intravitreal injections of Transebacillus for malignant thoracic or abdominal effusions, evaluated by changes in patient-reported outcome (PRO) scores before and after the intervention;
3-month puncture and/or drainage free rate; | 3 months
  an index to evaluate the efficacy of intrathecal injection in the treatment of malignant pleural or abdominal effusions for 3 months
6-month and 12-month OS rates | 1 year
  an index to evaluate the overall survival of intrathecal injection in the treatment of malignant pleural or abdominal effusions for 6 months or 12 months
Quality of Life score(EORTC QLQ-C30 ) | 1 year
  The quality of life consists of five function scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting), six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties), which will evaluate the score of life quality. The larger the score obtained, the worse the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xinxiang Medical university, Henan Province, China